CLINICAL TRIAL: NCT05109364
Title: The Effect of Alpha1- Adrenergic Receptor Antagonist Therapy on Cardiac and Striatal Transporter Uptake in Pre-Motor and Symptomatic Parkinson's Disease: a Follow Up Study
Brief Title: Terazosin and Parkinson's Disease Extension Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Michele Tagliati, MD, Professor and Vice Chairman, Director of Movement Disorders, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001770
Record Dates: First submitted 2021-10-13; First posted 2021-11-05 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Symptomatic Parkinson Disease; REM Sleep Behavior Disorder; Pre-motor Parkinson's Disease
Keywords: Parkinson's disease; REM sleep behavior disorder (RBD); Autonomic dysfunction; Neurodegeneration; Terazosin
MeSH Terms: conditions — Parkinson Disease, Secondary; REM Sleep Behavior Disorder; Parkinson Disease; Primary Dysautonomias; Nerve Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- terazosin therapy extension (Experimental): Primary procedures in this study are MIBG scan, DAT scan, NM-MRI, and terazosin medication. Subjects will return for research visits and imaging every six months for three years. The investigators hypothesize that the rate of decline in DAT scan123I-Ioflupane uptake will be slower in subjects who have received the alpha1- adrenergic receptor antagonist terazosin, resulting in a decreased clinical conversion rate to parkinsonism.
  Interventions: Drug: Terazosin therapy

INTERVENTIONS:
Drug: Terazosin therapy — Primary procedures in this study are MIBG scan, DAT scan, NM-MRI, and terazosin titration. Subjects will return for research visits and imaging every six months for three years. The investigators hypothesize that the rate of decline in DAT scan123I-Ioflupane uptake will be slower in subjects who have received the a1- Adrenergic Receptor Antagonist Terazosin, resulting in a decreased clinical conversion rate to parkinsonism.

SUMMARY:
The purpose of this study is to investigate the long-term effects of treatment with the selective post-synaptic a1-adrenergic blocker terazosin on serial in a population of subjects with defined pre-motor Parkinson's disease (PD) risks and abnormal imaging exams. Imaging changes will be correlated to the presence and severity of motor and non-motor symptoms of PD, measured by validated clinical scales and cardiac autonomic function tests.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the long-term effects of treatment with the selective post-synaptic a1-adrenergic blocker terazosin on serial 123 Ioflupane Dopamine Transporter single-photon emission-computed tomography (123I-FP DAT-SPECT) in a population of subjects with defined pre-motor PD risks (i.e., RBD and at least one among hyposmia, constipation, depression and color vision abnormality) and abnormal Iodine-123 meta-iodobenzylguanidine (123I-MIBG) uptake. Imaging changes will be correlated to the presence and severity of motor and non-motor symptoms of PD, measured by validated clinical scales and cardiac autonomic function tests. The rate of RBD clinical conversion to PD will be estimated and compared to available data in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the study "The Effect of alpha1- adrenergic receptor antagonist Therapy on Cardiac and Striatal Transporter Uptake in Pre-Motor and Symptomatic Parkinson's Disease" (STUDY #000540)
* Capacity to give informed consent

Exclusion Criteria:

* Secondary Parkinsonism, including tardive
* Concurrent dementia defined by a score lower than 22 on The Montreal Cognitive Assessment (MoCA)
* Concurrent severe depression defined by a Beck Depression Inventory-Fast Screen (BDI fast screen) score greater than 13
* Comorbidities related to sympathetic nervous system (SNS) hyperactivity
* Heart failure (LVEF <45%)
* Recent myocardial revascularization (<12 weeks)
* Hypertension (systolic blood pressure SBP>150mmHg (millimeters of mercury) or diastolic blood pressure DBP>100mmHg)
* Chronic Atrial fibrillation
* Concurrent Use of Beta-adrenergic antagonist
* Diabetes mellitus
* Chronic Obstructive Pulmonary Disease (COPD)
* Untreated Sever Sleep Apnea; Apnea-Hypopnea Index (AHI) > 30/h.
* Severely reduced kidney function (Glomerular Filtration Rate<30ml/min)
* Contraindications to the use of terazosin
* Recent myocardial infarction (<48 h)
* Ongoing angina pectoris
* Cardiogenic shock or prolonged hypotension
* Breast-feeding
* Current use of phosphodiesterase type 5 inhibitors: sildenafil (ViagraTM), tadalafil (CialisTM), or vardenafil (LevitraTM)
* History of priapism (persistent and painful erection)
* Neurogenic orthostatic hypotension defined as symptomatic decrease in BP > 20mmHg systolic or > 10mmHg diastolic and HR increase < 20bpm on supine to sitting or standing.
* Blood pressure less than 110 mm Hg systolic at screening or baseline visit
* Use of investigational drugs within 30 days before screening
* For female participant, pregnancy, or plans for child-bearing during study period
* Allergy/hypersensitivity to iodine or study medication

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in 123I-MIBG reuptake - early Heart to Mediastinal ratio (H/M) | Every 6 months for 3 years
  123I-MIBG early reuptake will be measured by Heart to Mediastinal ratio (H/M) which will be calculated from the early images after drawing regions of interest (7×7 pixels) over the upper mediastinum and circular ROI around the entire heart. MIBG abnormality cutoff will be set for values of late H/M <2.2.
Changes in 123I-MIBG reuptake - late Heart to Mediastinal ratio (H/M) | Every 6 months for 3 years
  123I-MIBG late reuptake will be measured by Heart to Mediastinal ratio (H/M) which will be calculated from the late images after drawing regions of interest (7×7 pixels) over the upper mediastinum and circular ROI around the entire heart. MIBG abnormality cutoff will be set for values of late H/M <2.2.
Changes in 123I-MIBG - Washout ratio (WR) | Every 6 months for 3 years
  123I-MIBG Washout ratio (WR) will be calculated using the following formula: [(early heart counts/pixel - early mediastinum counts/pixel) - (late heart counts/pixel decay-corrected - late mediastinum counts/pixel decay-corrected)]/(early heart counts/pixel - early mediastinum counts/pixel). Care will be taken to exclude lung or liver from the myocardial and large vessels and lung from the mediastinum region of interest. MIBG abnormality cutoff will be set for values of WR >30%.

SECONDARY OUTCOMES:
Diagnosis of PD or other synucleinopathies by the end of 3 years in the study population | 3 years
  Diagnosis of PD will be defined or ruled out according to the United Kingdom Parkinson's Disease Society Brain Bank (UKPDSBB) criteria
Changes in 123I-Ioflupane uptake | Every year for three years
  Measured by 123I-Ioflupane uptake, between baseline, year one, year two and year three.
Sensitivity and specificity of DAT Scan compared to MIBG in predicting RBD conversion to PD/other synucleinopathies | 3 years
  Integrity of pigmented neurons of substantia nigra.
Heart Rate Variability Analysis (HRV) compared to MIBG results in predicting RBD conversion to PD/other synucleinopathies | Every 6 months for 3 years
  Beat-to-beat intervals will be registered to assess sympatho-vagal balance. This measurement will be used for HRV analysis.

OTHER OUTCOMES:
MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III changes from without (OFF) medication between baseline and every 6 months for three years | Every 6 months for 3 years
  The Movement disorder society-unified Parkinson's disease rating scale (MDS-UPDRS) Part III will be administered at baseline and 26 weeks after study medication titration. Each item of the MDS-UPDRS has a possible rating from 0 to 4, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe.Clinical scales will be performed without (OFF) medication in those subjects that might be receiving dopaminergic drugs
Non-Motor Symptoms Scale (NMSS) changes between baseline and every 6 months for three years | Every 6 months for 3 years
  The NMSS measures non-motor symptoms over the previous month. Each symptom is scored with respect to: Severity: 0 = None, 1 = Mild; 2 = Moderate; 3 = Severe and Frequency: 1 = Rarely (<1/wk); 2 = Often (1/wk); 3 = Frequent (several times per week); 4 = Very Frequent (daily or all the time).
Scales for Outcomes in Parkinson's Disease - Autonomic Dysfunction (SCOPA-AUT) changes between baseline and every 6 months for three years | Every 6 months for 3 years
  The SCOPA-AUT was developed to evaluate autonomic symptoms in patients with Parkinson's disease. The scale is self-completed by patients and consists of 25 items assessing the following domains: gastrointestinal (7), urinary (6), cardiovascular (3), thermoregulatory (4), pupillomotor (1), and sexual (2 items for men and 2 items for women).
Rapid Eyes Movement (REM) sleep Behavior Disorder Screening questionnaire (RBDSQ) changes between baseline and every 6 months for three years | Every 6 months for 3 years
  The RBDSQ is a 10-item, patient self-rating instrument assessing the subject's sleep behavior with short questions that have to be answered by either "yes" or "no" that address frequency and content of dreams, their relationship to nocturnal movements/behavior, injuries of the bed partner, nocturnal vocalization, etc. The maximum total score of the RBDSQ is 13 points.
Smell changes as measured by University of Pennsylvania Smell Identification Test (UPSIT) | Every 6 months for 3 years
  University of Pennsylvania Smell Identification Test (UPSIT) changes.
Functional constipation score changes between baseline and every 6 months for three years | Every 6 months for 3 years
  Functional constipation will be assessed at screening and at 26 weeks after study medication titration using a questionnaire based on modified The Rome III Criteria for Functional Digestive Disorders (ROME III diagnostic criteria), which focuses on symptoms including straining, lumpy or hard stools, sensation of incomplete evacuation, sensation of anorectal obstruction or blockage, manual maneuvers to facilitate evacuation, and two or fewer bowel movements per week. This questionnaire is based on a six item self-report measures with a three point summated rating scale. The total score has a range of 0 to 12, with scores > 4 identifying functional constipation.
Color vision changes, as assessed using Hardy, Rand and Rittler (HRR) pseudoisochromatic Plates, between baseline and every 6 months for three years | Every 6 months for 3 years
  Color vision changes will be assessed using HRR pseudoisochromatic Plates.
Central insulin resistance changes between baseline and every 6 months for three years | Every 6 months for 3 years
  Measures of insulin sensitivity in neuronal-origin enriched plasma extracellular vesicles EVs (central IR) will be used to test the association of changes in such sensitivity to changes in MIBG uptake and clinical scores. For that purpose, plasma samples will be collected and stored and -80oC (celsius degrees) to allow for isolation of neuronal origin EVs at the completion of the study.
Differences in integrity of pigmented neurons in the locus coeruleus and substantia nigra between baseline, year one, year two and year three | 3 years
  This outcome will be measured by the content of neuromelanin, a product of catecholamine metabolism in locus coeruleus (LC) and substantia nigra (SN).
Correlation between changes in integrity of pigmented neurons of substantia nigra as measured by neuromelanin-sensitive magnetic resonance imaging (MRI) and 123I-Ioflupane uptake as measured by Dopamine Transporter Imaging (DAT scan) | 3 years
  These measurements will be aggregated to calculate the correlation between changes in neuromelanin content as measured by NM-MRI and dopamine content as measured by DAT scan
Heart Rate Variability (HRV) changes between baseline and every 6 months for three years | Every 6 months for 3 years
  Beat-to-beat intervals will be registered to assess sympatho-vagal balance. This measurement will be used for HRV analysis.
Peripheral insulin resistance (IR) changes between baseline and every 6 months for three years. | Every 6 months for 3 years
  Peripheral IR will be defined by the homeostasis model assessment of IR (HOMA-IR) defined as fasting glucose (mmol/L) x fasting insulin (mU/mL)/22.5. A cutoff HOMA index of 2.0, equivalent to <50% sensitivity, will be used to define IR. Subjects will be considered to have IR if they either have a HOMA≥2.0 and/or HbA1c≥5.7

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tagliati, MD, FAAN, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Academy of Sleep Medicine. International classification of sleep disor- ders 2nd ed.: Diagnostic and coding manual. Westchester, IL: American Academy of Sleep Medicine; 2005.
- [Background] Amino T, Orimo S, Itoh Y, Takahashi A, Uchihara T, Mizusawa H. Profound cardiac sympathetic denervation occurs in Parkinson disease. Brain Pathol. 2005 Jan;15(1):29-34. doi: 10.1111/j.1750-3639.2005.tb00097.x. PMID 15779234
- [Background] Boeve BF. REM sleep behavior disorder: Updated review of the core features, the REM sleep behavior disorder-neurodegenerative disease association, evolving concepts, controversies, and future directions. Ann N Y Acad Sci. 2010 Jan;1184:15-54. doi: 10.1111/j.1749-6632.2009.05115.x. PMID 20146689
- [Background] Braak H, Del Tredici K, Rub U, de Vos RA, Jansen Steur EN, Braak E. Staging of brain pathology related to sporadic Parkinson's disease. Neurobiol Aging. 2003 Mar-Apr;24(2):197-211. doi: 10.1016/s0197-4580(02)00065-9. PMID 12498954
- [Background] Cai R, Zhang Y, Simmering JE, Schultz JL, Li Y, Fernandez-Carasa I, Consiglio A, Raya A, Polgreen PM, Narayanan NS, Yuan Y, Chen Z, Su W, Han Y, Zhao C, Gao L, Ji X, Welsh MJ, Liu L. Enhancing glycolysis attenuates Parkinson's disease progression in models and clinical databases. J Clin Invest. 2019 Oct 1;129(10):4539-4549. doi: 10.1172/JCI129987. PMID 31524631
- [Background] Cedarbaum JM, Aghajanian GK. Catecholamine receptors on locus coeruleus neurons: pharmacological characterization. Eur J Pharmacol. 1977 Aug 15;44(4):375-85. doi: 10.1016/0014-2999(77)90312-0. No abstract available. PMID 330174
- [Background] Chang EB, Leung PS. Gastrintestinal Motility. In 'The Gastrointestinal System: Gastrointestinal, Nutritional and Hepatobiliary Physiology' P.S. Leung (ed.), Springer Science, Dordrecht 2014, 35-62.
- [Background] Clewett DV, Lee TH, Greening S, Ponzio A, Margalit E, Mather M. Neuromelanin marks the spot: identifying a locus coeruleus biomarker of cognitive reserve in healthy aging. Neurobiol Aging. 2016 Jan;37:117-126. doi: 10.1016/j.neurobiolaging.2015.09.019. Epub 2015 Oct 29. PMID 26521135
- [Background] de Milliano PA, van Eck-Smit BL, de Groot AC, Lie KI. Metoprolol-induced changes in myocardial (123)I-metaiodobenzylguanidine uptake in Parkinson's disease. Circulation. 2000 Nov 14;102(20):2553-4. doi: 10.1161/01.cir.102.20.2553. No abstract available. PMID 11076832
- [Background] de Peuter OR, Verberne HJ, Kok WE, van den Bogaard B, Schaap MC, Nieuwland R, Meijers JC, Somsen GA, Bakx A, Kamphuisen PW. Differential effects of nonselective versus selective beta-blockers on cardiac sympathetic activity and hemostasis in patients with heart failure. J Nucl Med. 2013 Oct;54(10):1733-9. doi: 10.2967/jnumed.113.120477. Epub 2013 Aug 22. PMID 23970363
- [Background] Dinan TG, Cryan JF. Regulation of the stress response by the gut microbiota: implications for psychoneuroendocrinology. Psychoneuroendocrinology. 2012 Sep;37(9):1369-78. doi: 10.1016/j.psyneuen.2012.03.007. Epub 2012 Apr 5. PMID 22483040
- [Background] Dorschner J, Farmakis G, Behnke S, Hellwig D, Schneider S, Fassbender K, Kirsch CM, Dillmann U, Spiegel J. Myocardial MIBG scintigraphy may predict the course of motor symptoms in Parkinson's disease. Parkinsonism Relat Disord. 2011 Jun;17(5):372-5. doi: 10.1016/j.parkreldis.2011.03.001. Epub 2011 Mar 21. PMID 21421334
- [Background] Fereshtehnejad SM, Montplaisir JY, Pelletier A, Gagnon JF, Berg D, Postuma RB. Validation of the MDS research criteria for prodromal Parkinson's disease: Longitudinal assessment in a REM sleep behavior disorder (RBD) cohort. Mov Disord. 2017 Jun;32(6):865-873. doi: 10.1002/mds.26989. Epub 2017 Apr 21. PMID 28429825
- [Background] Goldstein DS, Holmes C, Li ST, Bruce S, Metman LV, Cannon RO 3rd. Cardiac sympathetic denervation in Parkinson disease. Ann Intern Med. 2000 Sep 5;133(5):338-47. doi: 10.7326/0003-4819-133-5-200009050-00009. PMID 10979878
- [Background] Gronich N, Abernethy DR, Auriel E, Lavi I, Rennert G, Saliba W. beta2-adrenoceptor agonists and antagonists and risk of Parkinson's disease. Mov Disord. 2018 Sep;33(9):1465-1471. doi: 10.1002/mds.108. PMID 30311974
- [Background] Halsband C, Zapf A, Sixel-Doring F, Trenkwalder C, Mollenhauer B. The REM Sleep Behavior Disorder Screening Questionnaire is not Valid in De Novo Parkinson's Disease. Mov Disord Clin Pract. 2018 Mar 1;5(2):171-176. doi: 10.1002/mdc3.12591. eCollection 2018 Mar-Apr. PMID 30009211
- [Background] He SC, Niu Q. Subclinical neurophysiological effects of manganese in welding workers. Int J Immunopathol Pharmacol. 2004 May-Aug;17(2 Suppl):11-6. doi: 10.1177/03946320040170S203. PMID 15345186
- [Background] Heffernan DS, Inaba K, Arbabi S, Cotton BA. Sympathetic hyperactivity after traumatic brain injury and the role of beta-blocker therapy. J Trauma. 2010 Dec;69(6):1602-9. doi: 10.1097/TA.0b013e3181f2d3e8. No abstract available. PMID 21045744
- [Background] Hogg E, Athreya K, Basile C, Tan EE, Kaminski J, Tagliati M. High Prevalence of Undiagnosed Insulin Resistance in Non-Diabetic Subjects with Parkinson's Disease. J Parkinsons Dis. 2018;8(2):259-265. doi: 10.3233/JPD-181305. PMID 29614702
- [Background] Hughes KC, Gao X, Baker JM, Stephen C, Kim IY, Valeri L, Schwarzschild MA, Ascherio A. Non-motor features of Parkinson's disease in a nested case-control study of US men. J Neurol Neurosurg Psychiatry. 2018 Dec;89(12):1288-1295. doi: 10.1136/jnnp-2018-318275. Epub 2018 Aug 3. PMID 30076266
- [Background] Iranzo A, Santamaria J. Bisoprolol-induced rapid eye movement sleep behavior disorder. Am J Med. 1999 Oct;107(4):390-2. doi: 10.1016/s0002-9343(99)00245-4. No abstract available. PMID 10527042
- [Background] Iranzo A, Valldeoriola F, Lomena F, Molinuevo JL, Serradell M, Salamero M, Cot A, Ros D, Pavia J, Santamaria J, Tolosa E. Serial dopamine transporter imaging of nigrostriatal function in patients with idiopathic rapid-eye-movement sleep behaviour disorder: a prospective study. Lancet Neurol. 2011 Sep;10(9):797-805. doi: 10.1016/S1474-4422(11)70152-1. Epub 2011 Jul 28. PMID 21802993
- [Background] Iranzo A, Tolosa E, Gelpi E, Molinuevo JL, Valldeoriola F, Serradell M, Sanchez-Valle R, Vilaseca I, Lomena F, Vilas D, Llado A, Gaig C, Santamaria J. Neurodegenerative disease status and post-mortem pathology in idiopathic rapid-eye-movement sleep behaviour disorder: an observational cohort study. Lancet Neurol. 2013 May;12(5):443-53. doi: 10.1016/S1474-4422(13)70056-5. Epub 2013 Apr 3. PMID 23562390
- [Background] Iranzo A, Lomena F, Stockner H, Valldeoriola F, Vilaseca I, Salamero M, Molinuevo JL, Serradell M, Duch J, Pavia J, Gallego J, Seppi K, Hogl B, Tolosa E, Poewe W, Santamaria J; Sleep Innsbruck Barcelona (SINBAR) group. Decreased striatal dopamine transporter uptake and substantia nigra hyperechogenicity as risk markers of synucleinopathy in patients with idiopathic rapid-eye-movement sleep behaviour disorder: a prospective study [corrected]. Lancet Neurol. 2010 Nov;9(11):1070-7. doi: 10.1016/S1474-4422(10)70216-7. Epub 2010 Sep 16. PMID 20846908
- [Background] Iwanaga K, Wakabayashi K, Yoshimoto M, Tomita I, Satoh H, Takashima H, Satoh A, Seto M, Tsujihata M, Takahashi H. Lewy body-type degeneration in cardiac plexus in Parkinson's and incidental Lewy body diseases. Neurology. 1999 Apr 12;52(6):1269-71. doi: 10.1212/wnl.52.6.1269. PMID 10214756
- [Background] Jacob S, Rett K, Wicklmayr M, Agrawal B, Augustin HJ, Dietze GJ. Differential effect of chronic treatment with two beta-blocking agents on insulin sensitivity: the carvedilol-metoprolol study. J Hypertens. 1996 Apr;14(4):489-94. PMID 8761899
- [Background] Jacobson AF, Senior R, Cerqueira MD, Wong ND, Thomas GS, Lopez VA, Agostini D, Weiland F, Chandna H, Narula J; ADMIRE-HF Investigators. Myocardial iodine-123 meta-iodobenzylguanidine imaging and cardiac events in heart failure. Results of the prospective ADMIRE-HF (AdreView Myocardial Imaging for Risk Evaluation in Heart Failure) study. J Am Coll Cardiol. 2010 May 18;55(20):2212-21. doi: 10.1016/j.jacc.2010.01.014. Epub 2010 Feb 25. PMID 20188504
- [Background] Johnson ME, Stecher B, Labrie V, Brundin L, Brundin P. Triggers, Facilitators, and Aggravators: Redefining Parkinson's Disease Pathogenesis. Trends Neurosci. 2019 Jan;42(1):4-13. doi: 10.1016/j.tins.2018.09.007. Epub 2018 Oct 17. PMID 30342839
- [Background] Joyner MJ, Barnes JN, Hart EC, Wallin BG, Charkoudian N. Neural control of the circulation: how sex and age differences interact in humans. Compr Physiol. 2015 Jan;5(1):193-215. doi: 10.1002/cphy.c140005. PMID 25589269
- [Background] Keating GM, Jarvis B. Carvedilol: a review of its use in chronic heart failure. Drugs. 2003;63(16):1697-741. doi: 10.2165/00003495-200363160-00006. PMID 12904089
- [Background] Keren NI, Taheri S, Vazey EM, Morgan PS, Granholm AC, Aston-Jones GS, Eckert MA. Histologic validation of locus coeruleus MRI contrast in post-mortem tissue. Neuroimage. 2015 Jun;113:235-45. doi: 10.1016/j.neuroimage.2015.03.020. Epub 2015 Mar 17. PMID 25791783
- [Background] Knudsen K, Fedorova TD, Hansen AK, Sommerauer M, Otto M, Svendsen KB, Nahimi A, Stokholm MG, Pavese N, Beier CP, Brooks DJ, Borghammer P. In-vivo staging of pathology in REM sleep behaviour disorder: a multimodality imaging case-control study. Lancet Neurol. 2018 Jul;17(7):618-628. doi: 10.1016/S1474-4422(18)30162-5. Epub 2018 Jun 1. PMID 29866443
- [Background] Langston JW, Wiley JC, Tagliati M. Optimizing Parkinson's disease diagnosis: the role of a dual nuclear imaging algorithm. NPJ Parkinsons Dis. 2018 Feb 23;4:5. doi: 10.1038/s41531-018-0041-9. eCollection 2018. PMID 29507872
- [Background] Lotsch J, Daiker H, Hahner A, Ultsch A, Hummel T. Drug-target based cross-sectional analysis of olfactory drug effects. Eur J Clin Pharmacol. 2015 Apr;71(4):461-71. doi: 10.1007/s00228-015-1814-2. Epub 2015 Feb 11. PMID 25666029
- [Background] Mann DM, Yates PO. Lipoprotein pigments--their relationship to ageing in the human nervous system. II. The melanin content of pigmented nerve cells. Brain. 1974 Sep;97(3):489-98. doi: 10.1093/brain/97.1.489. No abstract available. PMID 4423478
- [Background] Marek KL, Seibyl JP, Zoghbi SS, Zea-Ponce Y, Baldwin RM, Fussell B, Charney DS, van Dyck C, Hoffer PB, Innis RP. [123I] beta-CIT/SPECT imaging demonstrates bilateral loss of dopamine transporters in hemi-Parkinson's disease. Neurology. 1996 Jan;46(1):231-7. doi: 10.1212/wnl.46.1.231. PMID 8559382
- [Background] Martinelli N, Olivieri O, Girelli D. Air particulate matter and cardiovascular disease: a narrative review. Eur J Intern Med. 2013 Jun;24(4):295-302. doi: 10.1016/j.ejim.2013.04.001. Epub 2013 May 4. PMID 23647842
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Mitsui J, Saito Y, Momose T, Shimizu J, Arai N, Shibahara J, Ugawa Y, Kanazawa I, Tsuji S, Murayama S. Pathology of the sympathetic nervous system corresponding to the decreased cardiac uptake in 123I-metaiodobenzylguanidine (MIBG) scintigraphy in a patient with Parkinson disease. J Neurol Sci. 2006 Apr 15;243(1-2):101-4. doi: 10.1016/j.jns.2005.11.034. Epub 2006 Jan 27. PMID 16442563
- [Background] Miyamoto T, Miyamoto M, Inoue Y, Usui Y, Suzuki K, Hirata K. Reduced cardiac 123I-MIBG scintigraphy in idiopathic REM sleep behavior disorder. Neurology. 2006 Dec 26;67(12):2236-8. doi: 10.1212/01.wnl.0000249313.25627.2e. PMID 17190953
- [Background] Mizutani Y, Nakamura T, Okada A, Suzuki J, Watanabe H, Hirayama M, Sobue G. Hyposmia and cardiovascular dysautonomia correlatively appear in early-stage Parkinson's disease. Parkinsonism Relat Disord. 2014 May;20(5):520-4. doi: 10.1016/j.parkreldis.2014.02.010. Epub 2014 Feb 20. PMID 24637128
- [Background] Morrison I, Frangulyan R, Riha RL. Beta-blockers as a cause of violent rapid eye movement sleep behavior disorder: a poorly recognized but common cause of violent parasomnias. Am J Med. 2011 Jan;124(1):e11. doi: 10.1016/j.amjmed.2010.04.023. Epub 2010 Sep 29. No abstract available. PMID 20887968
- [Background] Nakajo M, Shapiro B, Glowniak J, Sisson JC, Beierwaltes WH. Inverse relationship between cardiac accumulation of meta-[131I]iodobenzylguanidine (I-131 MIBG) and circulating catecholamines in suspected pheochromocytoma. J Nucl Med. 1983 Dec;24(12):1127-34. PMID 6644373
- [Background] Nomura T, Inoue Y, Kagimura T, Uemura Y, Nakashima K. Utility of the REM sleep behavior disorder screening questionnaire (RBDSQ) in Parkinson's disease patients. Sleep Med. 2011 Aug;12(7):711-3. doi: 10.1016/j.sleep.2011.01.015. Epub 2011 Jun 22. PMID 21700495
- [Background] Nul D, Zambrano C, Diaz A, Ferrante D, Varini S, Soifer S, Grancelli H, Doval H; Grupo de Estudio de la Sobrevida en la Insuficiencia Cardiaca en Argentina. Impact of a standardized titration protocol with carvedilol in heart failure: safety, tolerability, and efficacy-a report from the GESICA registry. Cardiovasc Drugs Ther. 2005 Mar;19(2):125-34. doi: 10.1007/s10557-005-1497-5. PMID 16025231
- [Background] Orimo S, Ozawa E, Nakade S, Sugimoto T, Mizusawa H. (123)I-metaiodobenzylguanidine myocardial scintigraphy in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1999 Aug;67(2):189-94. doi: 10.1136/jnnp.67.2.189. PMID 10406987
- [Background] Orimo S, Uchihara T, Nakamura A, Mori F, Kakita A, Wakabayashi K, Takahashi H. Axonal alpha-synuclein aggregates herald centripetal degeneration of cardiac sympathetic nerve in Parkinson's disease. Brain. 2008 Mar;131(Pt 3):642-50. doi: 10.1093/brain/awm302. Epub 2007 Dec 13. PMID 18079166
- [Background] Orimo S, Suzuki M, Inaba A, Mizusawa H. 123I-MIBG myocardial scintigraphy for differentiating Parkinson's disease from other neurodegenerative parkinsonism: a systematic review and meta-analysis. Parkinsonism Relat Disord. 2012 Jun;18(5):494-500. doi: 10.1016/j.parkreldis.2012.01.009. Epub 2012 Feb 8. PMID 22321865
- [Background] Otsuka N, Ohi M, Chin K, Kita H, Noguchi T, Hata T, Nohara R, Hosokawa R, Fujita M, Kuno K. Assessment of cardiac sympathetic function with iodine-123-MIBG imaging in obstructive sleep apnea syndrome. J Nucl Med. 1997 Apr;38(4):567-72. PMID 9098203
- [Background] Packer M, Bristow MR, Cohn JN, Colucci WS, Fowler MB, Gilbert EM, Shusterman NH. The effect of carvedilol on morbidity and mortality in patients with chronic heart failure. U.S. Carvedilol Heart Failure Study Group. N Engl J Med. 1996 May 23;334(21):1349-55. doi: 10.1056/NEJM199605233342101. PMID 8614419
- [Background] Pagano G, Tan EE, Haider JM, Bautista A, Tagliati M. Constipation is reduced by beta-blockers and increased by dopaminergic medications in Parkinson's disease. Parkinsonism Relat Disord. 2015 Feb;21(2):120-5. doi: 10.1016/j.parkreldis.2014.11.015. Epub 2014 Nov 25. PMID 25483722
- [Background] Postuma RB, Montplaisir J, Lanfranchi P, Blais H, Rompre S, Colombo R, Gagnon JF. Cardiac autonomic denervation in Parkinson's disease is linked to REM sleep behavior disorder. Mov Disord. 2011 Jul;26(8):1529-33. doi: 10.1002/mds.23677. Epub 2011 Apr 29. PMID 21538520
- [Background] Postuma RB, Aarsland D, Barone P, Burn DJ, Hawkes CH, Oertel W, Ziemssen T. Identifying prodromal Parkinson's disease: pre-motor disorders in Parkinson's disease. Mov Disord. 2012 Apr 15;27(5):617-26. doi: 10.1002/mds.24996. PMID 22508280
- [Background] Postuma RB, Gagnon JF, Bertrand JA, Genier Marchand D, Montplaisir JY. Parkinson risk in idiopathic REM sleep behavior disorder: preparing for neuroprotective trials. Neurology. 2015 Mar 17;84(11):1104-13. doi: 10.1212/WNL.0000000000001364. Epub 2015 Feb 13. PMID 25681454
- [Background] Pyatigorskaya N, Gaurav R, Arnaldi D, Leu-Semenescu S, Yahia-Cherif L, Valabregue R, Vidailhet M, Arnulf I, Lehericy S. Magnetic Resonance Imaging Biomarkers to Assess Substantia Nigra Damage in Idiopathic Rapid Eye Movement Sleep Behavior Disorder. Sleep. 2017 Nov 1;40(11). doi: 10.1093/sleep/zsx149. PMID 28958075
- [Background] Sakakibara R, Tateno F, Kishi M, Tsuyusaki Y, Terada H, Inaoka T. MIBG myocardial scintigraphy in pre-motor Parkinson's disease: a review. Parkinsonism Relat Disord. 2014 Mar;20(3):267-73. doi: 10.1016/j.parkreldis.2013.11.001. Epub 2013 Nov 21. PMID 24332912
- [Background] Sakata K, Shirotani M, Yoshida H, Kurata C. Cardiac sympathetic nervous system in early essential hypertension assessed by 123I-MIBG. J Nucl Med. 1999 Jan;40(1):6-11. PMID 9935049
- [Background] Sasaki M, Shibata E, Tohyama K, Takahashi J, Otsuka K, Tsuchiya K, Takahashi S, Ehara S, Terayama Y, Sakai A. Neuromelanin magnetic resonance imaging of locus ceruleus and substantia nigra in Parkinson's disease. Neuroreport. 2006 Jul 31;17(11):1215-8. doi: 10.1097/01.wnr.0000227984.84927.a7. PMID 16837857
- [Background] Scheer FA, Morris CJ, Garcia JI, Smales C, Kelly EE, Marks J, Malhotra A, Shea SA. Repeated melatonin supplementation improves sleep in hypertensive patients treated with beta-blockers: a randomized controlled trial. Sleep. 2012 Oct 1;35(10):1395-402. doi: 10.5665/sleep.2122. PMID 23024438
- [Background] Scott LA, Kench PL. Cardiac autonomic neuropathy in the diabetic patient: does 123I-MIBG imaging have a role to play in early diagnosis? J Nucl Med Technol. 2004 Jun;32(2):66-71. PMID 15175402
- [Background] Searles Nielsen S, Gross A, Camacho-Soto A, Willis AW, Racette BA. beta2-adrenoreceptor medications and risk of Parkinson disease. Ann Neurol. 2018 Nov;84(5):683-693. doi: 10.1002/ana.25341. Epub 2018 Oct 30. PMID 30225948
- [Background] Seravalle G, Piperno A, Mariani R, Pelloni I, Facchetti R, Dell'Oro R, Cuspidi C, Mancia G, Grassi G. Alterations in sympathetic nerve traffic in genetic haemochromatosis before and after iron depletion therapy: a microneurographic study. Eur Heart J. 2016 Mar 21;37(12):988-95. doi: 10.1093/eurheartj/ehv696. Epub 2015 Dec 28. PMID 26715163
- [Background] Schenck CH, Bundlie SR, Mahowald MW. Delayed emergence of a parkinsonian disorder in 38% of 29 older men initially diagnosed with idiopathic rapid eye movement sleep behaviour disorder. Neurology. 1996 Feb;46(2):388-93. doi: 10.1212/wnl.46.2.388. PMID 8614500
- [Background] Schenck CH, Boeve BF, Mahowald MW. Delayed emergence of a parkinsonian disorder or dementia in 81% of older men initially diagnosed with idiopathic rapid eye movement sleep behavior disorder: a 16-year update on a previously reported series. Sleep Med. 2013 Aug;14(8):744-8. doi: 10.1016/j.sleep.2012.10.009. Epub 2013 Jan 22. PMID 23347909
- [Background] Spiegel J, Mollers MO, Jost WH, Fuss G, Samnick S, Dillmann U, Becker G, Kirsch CM. FP-CIT and MIBG scintigraphy in early Parkinson's disease. Mov Disord. 2005 May;20(5):552-61. doi: 10.1002/mds.20369. PMID 15645531
- [Background] Spiegel J, Hellwig D, Samnick S, Jost W, Mollers MO, Fassbender K, Kirsch CM, Dillmann U. Striatal FP-CIT uptake differs in the subtypes of early Parkinson's disease. J Neural Transm (Vienna). 2007 Mar;114(3):331-5. doi: 10.1007/s00702-006-0518-2. Epub 2006 May 24. PMID 16715205
- [Background] Spiegel J, Hellwig D, Jost WH, Farmakis G, Samnick S, Fassbender K, Kirsch CM, Dillmann U. Cerebral and Extracranial Neurodegeneration are Strongly Coupled in Parkinson's Disease. Open Neurol J. 2007;1:1-4. doi: 10.2174/1874205X00701010001. Epub 2007 Aug 22. PMID 19018276
- [Background] Stoschitzky K, Koshucharova G, Lercher P, Maier R, Sakotnik A, Klein W, Liebmann PM, Lindner W. Stereoselective effects of (R)- and (S)-carvedilol in humans. Chirality. 2001 Jul;13(7):342-6. doi: 10.1002/chir.1042. PMID 11400186
- [Background] Taki J, Nakajima K, Hwang EH, Matsunari I, Komai K, Yoshita M, Sakajiri K, Tonami N. Peripheral sympathetic dysfunction in patients with Parkinson's disease without autonomic failure is heart selective and disease specific. taki@med.kanazawa-u.ac.jp. Eur J Nucl Med. 2000 May;27(5):566-73. doi: 10.1007/s002590050544. PMID 10853813
- [Background] Travin MI, Matsunari I, Thomas GS, Nakajima K, Yoshinaga K. How do we establish cardiac sympathetic nervous system imaging with 123I-mIBG in clinical practice? Perspectives and lessons from Japan and the US. J Nucl Cardiol. 2019 Aug;26(4):1434-1451. doi: 10.1007/s12350-018-1394-5. Epub 2018 Sep 3. PMID 30178272
- [Background] Treglia G, Stefanelli A, Bruno I, Giordano A. Clinical usefulness of myocardial innervation imaging using Iodine-123-meta-iodobenzylguanidine scintigraphy in evaluating the effectiveness of pharmacological treatments in patients with heart failure: an overview. Eur Rev Med Pharmacol Sci. 2013 Jan;17(1):56-68. PMID 23329524
- [Background] Valappil RA, Black JE, Broderick MJ, Carrillo O, Frenette E, Sullivan SS, Goldman SM, Tanner CM, Langston JW. Exploring the electrocardiogram as a potential tool to screen for premotor Parkinson's disease. Mov Disord. 2010 Oct 30;25(14):2296-303. doi: 10.1002/mds.23348. PMID 20976736
- [Background] Varrone A, Dickson JC, Tossici-Bolt L, Sera T, Asenbaum S, Booij J, Kapucu OL, Kluge A, Knudsen GM, Koulibaly PM, Nobili F, Pagani M, Sabri O, Vander Borght T, Van Laere K, Tatsch K. European multicentre database of healthy controls for [123I]FP-CIT SPECT (ENC-DAT): age-related effects, gender differences and evaluation of different methods of analysis. Eur J Nucl Med Mol Imaging. 2013 Jan;40(2):213-27. doi: 10.1007/s00259-012-2276-8. Epub 2012 Nov 16. PMID 23160999
- [Background] Velseboer DC, de Haan RJ, Wieling W, Goldstein DS, de Bie RM. Prevalence of orthostatic hypotension in Parkinson's disease: a systematic review and meta-analysis. Parkinsonism Relat Disord. 2011 Dec;17(10):724-9. doi: 10.1016/j.parkreldis.2011.04.016. Epub 2011 May 14. PMID 21571570
- [Background] Verberne HJ, Brewster LM, Somsen GA, van Eck-Smit BL. Prognostic value of myocardial 123I-metaiodobenzylguanidine (MIBG) parameters in patients with heart failure: a systematic review. Eur Heart J. 2008 May;29(9):1147-59. doi: 10.1093/eurheartj/ehn113. Epub 2008 Mar 17. PMID 18349024
- [Background] Wieland DM, Brown LE, Rogers WL, Worthington KC, Wu JL, Clinthorne NH, Otto CA, Swanson DP, Beierwaltes WH. Myocardial imaging with a radioiodinated norepinephrine storage analog. J Nucl Med. 1981 Jan;22(1):22-31. PMID 7452352
- [Background] Zecca L, Tampellini D, Gerlach M, Riederer P, Fariello RG, Sulzer D. Substantia nigra neuromelanin: structure, synthesis, and molecular behaviour. Mol Pathol. 2001 Dec;54(6):414-8. PMID 11724917
- [Background] Zimnik NC, Treadway T, Smith RS, Araneda RC. alpha(1A)-Adrenergic regulation of inhibition in the olfactory bulb. J Physiol. 2013 Apr 1;591(7):1631-43. doi: 10.1113/jphysiol.2012.248591. Epub 2012 Dec 24. PMID 23266935